CLINICAL TRIAL: NCT03315455
Title: A Randomized, Multicenter, Open-Label, Phase III Clinical Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of Prophylactic Emicizumab Versus No Prophylaxis in Hemophilia A Patients
Brief Title: Efficacy, Safety, and Pharmacokinetic Study of Prophylactic Emicizumab Versus No Prophylaxis in Hemophilia A Participants
Acronym: HAVEN 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO39309
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm C (Control): No Prophylaxis, Then Emicizumab (Active Comparator): Participants ≥12 years old with hemophilia A (with or without FVIII inhibitors) who are randomized to Arm C will not receive any prophylactic treatment for at least 24 weeks. After 24 weeks, participants will have the opportunity to switch to receive emicizumab prophylaxis at 3 mg/kg QW via SC injection for 4 weeks, followed by 6 mg/kg Q4W until marketing authorization as part of this study or a separate extension study, as long as they derive clinical benefit. Participants will continue to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
  Interventions: Drug: Emicizumab
- Arm A: Emicizumab Prophylaxis at 1.5 mg/kg QW (Experimental): Participants ≥12 years old with hemophilia A (with or without FVIII inhibitors) who are randomized to Arm A will receive prophylactic emicizumab at a dose of 3 mg/kg via SC injection QW for first 4 weeks, followed by 1.5 mg/kg via SC injection Q4W for at least 24 weeks. After 24 weeks treatment, participants will be allowed to continue emicizumab until marketing authorization as part of this study or a separate extension study, as long as they derive clinical benefit. Participants will continue to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
  Interventions: Drug: Emicizumab
- Arm B: Emicizumab Prophylaxis at 6 mg/kg Q4W (Experimental): Participants ≥12 years old with hemophilia A (with or without FVIII inhibitors) who are randomized to Arm B will receive prophylactic emicizumab at a dose of 3 mg/kg via SC injection QW for first 4 weeks, followed by 6 mg/kg via SC injection Q4W for at least 24 weeks. After 24 weeks treatment, participants will be allowed to continue emicizumab until marketing authorization as part of this study or a separate extension study, as long as they derive clinical benefit. Participants will continue to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
  Interventions: Drug: Emicizumab
- Arm D: Emicizumab Prophylaxis at 1.5 mg/kg QW (Experimental): Participants <12 years old with hemophilia A and FVIII inhibitors who are enrolled to Arm D will receive prophylactic emicizumab at a dose of 3 mg/kg via SC injection QW for first 4 weeks, followed by 1.5 mg/kg via SC injection QW for at least 24 weeks. After 24 weeks treatment, participants will be allowed to continue emicizumab until marketing authorization as part of this study or a separate extension study, as long as they derive clinical benefit. Participants will continue to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Emicizumab will be administered via subcutaneous (SC) injection, as described for each treatment arm.
  Other Names: Hemlibra; RO5534262; RG6013; ACE910

SUMMARY:
This multicenter, open-label, Phase 3 study with randomized and non-randomized arms is designed to investigate the efficacy, safety, and pharmacokinetics of emicizumab in participants with hemophilia A regardless of factor VIII (FVIII) inhibitor status. Participants greater than or equal to (≥)12 years old who received episodic therapy with FVIII or bypassing agents prior to study entry and experienced at least 5 bleeds over the prior 24 weeks will be randomized in a 2:2:1 ratio to the following regimens: Arm A: Emicizumab prophylaxis at 3 milligrams per kilogram (mg/kg) once every week (QW) subcutaneously (SC) for 4 weeks, followed by 1.5 mg/kg QW SC; Arm B: Emicizumab prophylaxis at 3 mg/kg QW SC for 4 weeks, followed by 6 mg/kg once every 4 weeks (Q4W) SC; and Arm C: No prophylaxis (control arm). In addition, pediatric participants less than (<)12 years old with hemophilia A and FVIII inhibitors who received episodic therapy with bypassing agents prior to study entry will be enrolled to Arm D: Emicizumab prophylaxis at 3 mg/kg QW SC for 4 weeks, followed by 1.5 mg/kg QW SC.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Arms A, B, and C:

* Diagnosis of severe congenital hemophilia A or hemophilia A with FVIII inhibitors
* Aged 12 years or older at the time of informed consent
* Body weight ≥40 kilograms (kg) at the time of screening
* Participants without FVIII inhibitors (<0.6 Bethesda unit per milliliter [BU/mL]) who completed successful immune tolerance induction (ITI) must have done so at least 5 years before screening and have no evidence of inhibitor recurrence (permanent or temporary)
* Documentation of the details of episodic therapy (FVIII or bypassing agents) and of number of bleeding episodes for at least the last 24 weeks and ≥5 bleeds in the last 24 weeks prior to study entry
* Adequate hematologic, hepatic, and renal function
* For women of child bearing potential: agreement to remain abstinent or use a protocol defined contraceptive measure during the treatment period and for at least 5 elimination half-lives (24 weeks) after the last dose of study drug

Inclusion Criteria for Arm D:

* Diagnosis of congenital hemophilia A of any severity and documented history of high-titer inhibitor (i.e., ≥5 BU/mL)
* Children <12 years old at time of informed consent
* Body weight >3 kg at time of informed consent
* Requires treatment with bypassing agents
* Adequate hematologic, hepatic, and renal function
* For female participants who are of childbearing potential, follow the same contraception criteria as listed above for Arms A, B, and C

Exclusion Criteria:

Exclusion Criteria for Arms A, B, and C:

* Inherited or acquired bleeding disorder other than hemophilia A
* At high risk for thrombotic microangiopathy, in the investigator's judgment
* History of illicit drug or alcohol abuse within 48 weeks prior to screening, in the investigator's judgment
* Previous (in the past 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease
* Other conditions that may increase risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Known human immuno-deficiency virus (HIV) infection with cluster of differentiation 4 (CD4) count <200 cells/microliter (cells/mcL) within 24 weeks prior to screening. Participants with HIV infection who have CD4 >200 cells/mcL and meet all other criteria are eligible
* Use of systemic immunomodulators at enrollment or planned use during the study, with the exception of anti-retroviral therapy
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose additional risk, or would, in the opinion of the investigator, preclude the participant's safe participation in and completion of the study
* Planned surgery (excluding minor procedures such as tooth extraction or incision and drainage) during the study
* Receipt of: Emicizumab in a prior investigational study; An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration; A non-hemophilia-related investigational drug concurrently, within last 30 days or 5 half-lives, whichever is shorter
* Pregnant or lactating, or intending to become pregnant during the study

Exclusion Criteria for Arm D:

* Inherited or acquired bleeding disorder other than hemophilia A
* Ongoing (or plan to receive during the study) ITI therapy or prophylaxis treatment with FVIII
* Previous (in the past 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease
* Other diseases that may increase risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Known infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV)
* At high risk for thrombotic microangiopathy, in the investigator's judgment
* Use of systemic immunomodulators at enrollment or planned use during the study
* Planned surgery (excluding minor procedures such as tooth extraction or incision and drainage) during the study
* Inability (or unwillingness by caregiver) to receive (allow receipt of) blood or blood products (or any standard-of-care treatment for a life-threatening condition)
* Receipt of: Emicizumab in a prior investigational study; An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration; A non-hemophilia-related investigational drug concurrently, within last 30 days or 5 half-lives, whichever is shorter
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose additional risk, or would, in the opinion of the investigator, preclude the participant's safe participation in and completion of the study
* Pregnant or lactating, or intending to become pregnant during the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2025-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- China (7):
  - Peking Union Medical College Hospital, Beijing
  - Xiangya Hospital of Centre-South University, Changsha
  - Southern Medical University Nanfang Hospital, Guangdong Province Guangzhou City
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Tianjin Institute of Hematology & Blood Diseases Hospital, Tianjin
  - Xiehe Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Malaysia (2):
  - Penang General Hospital, George Town, Pulau Pinang
  - Queen Elizabeth Hospital, Sabah, Sabah
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 76 patients were screened for eligibility, 6 of whom were deemed ineligible, and 70 participants were randomized to this study (Arms A, B, and C). Arm D was added later in a protocol amendment (Version 4) after the study had already started. For Arm D, a total of 16 patients were screened and 15 patients were enrolled.
Groups:
- Arm C: No Prophylaxis (Control), Then Emicizumab: Participants ≥12 years old with hemophilia A (with or without FVIII inhibitors) who were randomized to Arm C did not receive any prophylactic treatment for at least 24 weeks (Control). After 24 weeks, participants had the opportunity to switch to receive emicizumab prophylaxis at 3 mg/kg QW via SC injection for 4 weeks, followed by 6 mg/kg Q4W until marketing authorization, as part of this study or a separate extension study, as long as they derived clinical benefit. Participants continued to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
- Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW: Participants ≥12 years old with hemophilia A (with or without FVIII inhibitors) who were randomized to Arm A received prophylactic emicizumab at a dose of 3 mg/kg via SC injection QW for the first 4 weeks, followed by 1.5 mg/kg via SC injection QW for at least 24 weeks. After 24 weeks of treatment, participants were allowed to continue receiving emicizumab until marketing authorization, as part of this study or a separate extension study, as long as they derived clinical benefit. Participants continued to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
- Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W: Participants ≥12 years old with hemophilia A (with or without FVIII inhibitors) who were randomized to Arm B received prophylactic emicizumab at a dose of 3 mg/kg via SC injection QW for the first 4 weeks, followed by 6 mg/kg via SC injection Q4W for at least 24 weeks. After 24 weeks of treatment, participants were allowed to continue receiving emicizumab until marketing authorization, as part of this study or a separate extension study, as long as they derived clinical benefit. Participants continued to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
- Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW: Participants <12 years old with hemophilia A and FVIII inhibitors who were enrolled to Arm D received prophylactic emicizumab at a dose of 3 mg/kg via SC injection QW for the first 4 weeks, followed by 1.5 mg/kg via SC injection QW for at least 24 weeks. After 24 weeks of treatment, participants were allowed to continue receiving emicizumab until marketing authorization, as part of this study or a separate extension study, as long as they derived clinical benefit. Participants continued to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
Period: Overall Study
Arm/Group | Arm C: No Prophylaxis (Control), Then Emicizumab | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Started | 14 | 29 | 27 | 15
Completed 24 Weeks in the Study | 14 (After completing 24 weeks of no prophylaxis, all participants in Arm C switched to receive emicizumab (Arm C emi).) | 29 | 27 | 15
Completed | 1 | 4 | 10 | 0
Not Completed | 13 | 25 | 17 | 15
Not completed — Ongoing in the Study | 13 | 24 | 17 | 15
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm C: No Prophylaxis (Control), Then Emicizumab | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW | Total
Number analyzed (Participants) | 14 | 29 | 27 | 15 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.5 (10.9) | 32.2 (12.0) | 28.6 (13.5) | 7.5 (2.2) | 25.9 (14.2)
Age, Customized [Count of Participants; unit: Participants]
  <18 Years Old | 2 | 3 | 6 | 15 | 26
  ≥18 to <65 Years Old | 12 | 26 | 20 | 0 | 58
  ≥65 Years Old | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 14 | 29 | 27 | 15 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 14 | 29 | 27 | 15 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 14 | 29 | 27 | 15 | 85
Factor VIII (FVIII) Inhibitor Status at Study Entry [Count of Participants; unit: Participants]
  FVIII Inhibitor Positive | 3 | 5 | 7 | 15 | 30
  FVIII Inhibitor Negative (Non-Inhibitor) | 11 | 24 | 20 | 0 | 55
Categorical Number of Bleeds (<9 or ≥9) in the Past 24 Weeks Prior to Study Entry [Count of Participants; unit: Participants]
  <9 Bleeds | 3 | 7 | 6 | 5 | 21
  ≥9 Bleeds | 11 | 22 | 21 | 10 | 64

OUTCOME MEASURES:

1. Primary Outcome: Model-Based Annualized Bleeding Rate for Treated Bleeds
Description: The number of treated bleeds over the efficacy period was estimated as an annualized bleeding rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated bleed was defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: Treated bleeds per year
Groups:
- Arm C (Control): No Prophylaxis: Participants ≥12 years old with hemophilia A (with or without FVIII inhibitors) who were randomized to Arm C did not receive any prophylactic treatment for the first 24 weeks of the study (Control). Participants continued to receive standard-of-care treatments on an episodic basis for the treatment of bleeds during the study.
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated bleeds per year | 27.0 [13.29 to 54.91] | 1.0 [0.53 to 1.85] | 1.0 [0.50 to 1.84] | 1.2 [0.48 to 3.13]
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW; H0 (null hypothesis): ABR Ratio = 1; versus, H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — Statistical significance was controlled at a 2-sided alpha level of 0.05. Hierarchical testing was used to account for multiple comparisons; ABR Ratio = 0.04, 95% CI 2-sided [0.016 to 0.084] — The ABR ratio was calculated as Arm A vs. Arm C
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W; H0 (null hypothesis): ABR Ratio = 1; versus, H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.04, 95% CI 2-sided [0.015 to 0.082] — The ABR ratio was calculated as Arm B vs. Arm C

2. Primary Outcome: Mean Calculated Annualized Bleeding Rate for Treated Bleeds
Description: The number of treated bleeds over the efficacy period is presented here as a calculated annualized bleeding rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated bleed was defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Mean (95% Confidence Interval); unit: Treated bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated bleeds per year | 43.7 [31.71 to 58.71] | 1.4 [0.09 to 6.29] | 1.5 [0.10 to 6.38] | 1.2 [0.05 to 5.94]

3. Primary Outcome: Median Calculated Annualized Bleeding Rate for Treated Bleeds
Description: as for outcome 2
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Median (Inter-Quartile Range); unit: Treated bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated bleeds per year | 45.3 [21.74 to 70.49] | 0.0 [0.00 to 1.23] | 0.0 [0.00 to 2.26] | 0.0 [0.00 to 2.08]

4. Secondary Outcome: Model-Based Annualized Bleeding Rate for All Bleeds
Description: The number of all bleeds over the efficacy period was estimated as an annualized bleeding rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule meant that two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: All bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
All bleeds per year | 41.1 [26.37 to 64.19] | 1.9 [1.23 to 2.97] | 2.1 [1.33 to 3.26] | 3.8 [2.21 to 6.69]
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW; H0 (null hypothesis): ABR Ratio = 1; versus, H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.05, 95% CI 2-sided [0.026 to 0.084] — The ABR ratio was calculated as Arm A vs. Arm C
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W; H0 (null hypothesis): ABR Ratio = 1; versus, H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.05, 95% CI 2-sided [0.028 to 0.092] — The ABR ratio was calculated as Arm B vs. Arm C

5. Secondary Outcome: Mean Calculated Annualized Bleeding Rate for All Bleeds
Description: The number of all bleeds over the efficacy period is presented here as a calculated annualized bleeding rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule meant that two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Mean (95% Confidence Interval); unit: All bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
All bleeds per year | 53.0 [39.71 to 69.33] | 2.7 [0.51 to 8.37] | 3.1 [0.67 to 8.94] | 3.8 [1.01 to 10.01]

6. Secondary Outcome: Median Calculated Annualized Bleeding Rate for All Bleeds
Description: as for outcome 5
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Median (Inter-Quartile Range); unit: All bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
All bleeds per year | 56.7 [26.09 to 70.81] | 1.5 [0.00 to 4.21] | 1.9 [0.00 to 5.62] | 2.1 [0.00 to 5.77]

7. Secondary Outcome: Model-Based Annualized Bleeding Rate for Treated Spontaneous Bleeds
Description: The number of treated spontaneous bleeds over the efficacy period was estimated as an annualized bleeding rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated spontaneous bleed was defined as a treated bleed (bleed directly followed by a hemophilia medication reported to be a "treatment for bleed") with no other known contributing factor such as trauma or procedure/surgery. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: Treated spontaneous bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated spontaneous bleeds per year | 23.6 [9.28 to 60.03] | 0.4 [0.18 to 0.96] | 0.5 [0.20 to 1.12] | 0.6 [0.18 to 2.16]
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW; H0 (null hypothesis): ABR Ratio = 1; versus, H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.02, 95% CI 2-sided [0.006 to 0.053] — The ABR ratio was calculated as Arm A vs. Arm C
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W; H0 (null hypothesis): ABR Ratio = 1; versus, H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.02, 95% CI 2-sided [0.007 to 0.059] — The ABR ratio was calculated as Arm B vs. Arm C

8. Secondary Outcome: Mean Calculated Annualized Bleeding Rate for Treated Spontaneous Bleeds
Description: The number of treated spontaneous bleeds over the efficacy period is presented here as a calculated annualized bleeding rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated spontaneous bleed was defined as a treated bleed (bleed directly followed by a hemophilia medication reported to be a "treatment for bleed") with no other known contributing factor such as trauma or procedure/surgery. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Mean (95% Confidence Interval); unit: Treated spontaneous bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated spontaneous bleeds per year | 30.9 [20.95 to 43.85] | 0.5 [0.00 to 4.66] | 0.6 [0.00 to 4.88] | 0.6 [0.00 to 4.92]

9. Secondary Outcome: Median Calculated Annualized Bleeding Rate for Treated Spontaneous Bleeds
Description: as for outcome 8
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Median (Inter-Quartile Range); unit: Treated spontaneous bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated spontaneous bleeds per year | 21.8 [6.48 to 52.18] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.96] | 0.0 [0.00 to 0.00]

10. Secondary Outcome: Model-Based Annualized Bleeding Rate for Treated Joint Bleeds
Description: The number of treated joint bleeds over the efficacy period was estimated as an annualized bleeding rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated joint bleed was defined as a bleed with type reported as "joint" based on at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline, and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: Treated joint bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated joint bleeds per year | 17.7 [8.33 to 37.57] | 0.7 [0.36 to 1.46] | 0.6 [0.28 to 1.22] | 0.1 [0.02 to 0.88]
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW; H0 (null hypothesis): ABR Ratio = 1; versus, H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.04, 95% CI 2-sided [0.017 to 0.102] — The ABR ratio was calculated as Arm A vs. Arm C
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W; H0 (null hypothesis): ABR Ratio = 1; versus, H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.03, 95% CI 2-sided [0.013 to 0.084] — The ABR ratio was calculated as Arm B vs. Arm C

11. Secondary Outcome: Mean Calculated Annualized Bleeding Rate for Treated Joint Bleeds
Description: The number of treated joint bleeds over the efficacy period is presented here as a calculated annualized bleeding rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated joint bleed was defined as a bleed with type reported as "joint" based on at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline, and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Mean (95% Confidence Interval); unit: Treated joint bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated joint bleeds per year | 25.5 [16.62 to 37.56] | 1.0 [0.02 to 5.57] | 0.8 [0.01 to 5.20] | 0.1 [0.00 to 3.93]

12. Secondary Outcome: Median Calculated Annualized Bleeding Rate for Treated Joint Bleeds
Description: as for outcome 11
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Median (Inter-Quartile Range); unit: Treated joint bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated joint bleeds per year | 10.9 [8.70 to 50.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 1.40] | 0.0 [0.00 to 0.00]

13. Secondary Outcome: Model-Based Annualized Bleeding Rate for Treated Target Joint Bleeds
Description: The number of treated target joint bleeds over the efficacy period was estimated as an annualized bleeding rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated target joint bleed was defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry or an unresolved target joint (target joint that does not fulfil ≤2 bleeds into this joint within a consecutive 12-month period), and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: Treated target joint bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated target joint bleeds per year | 8.6 [3.15 to 23.42] | 0.4 [0.18 to 1.09] | 0.3 [0.12 to 0.85] | NA [NA to NA] — The model-based ABR was not estimable because too few events had occurred.
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW; Test type: Superiority; p < 0.0001, Stratified Wald test — Not controlled for Type I error; ABR Ratio = 0.05, 95% CI 2-sided [0.016 to 0.163] — The ABR ratio was calculated as Arm A vs. Arm C
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W; Test type: Superiority; p < 0.0001, ABR Ratio — Not controlled for Type I error; ABR Ratio = 0.04, 95% CI 2-sided [0.011 to 0.122] — The ABR ratio was calculated as Arm B vs. Arm C

14. Secondary Outcome: Mean Calculated Annualized Bleeding Rate for Treated Target Joint Bleeds
Description: The number of treated target joint bleeds over the efficacy period is presented here as a calculated annualized bleeding rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated target joint bleed was defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry or an unresolved target joint (target joint that does not fulfil ≤2 bleeds into this joint within a consecutive 12-month period), and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Mean (95% Confidence Interval); unit: Treated target joint bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated target joint bleeds per year | 15.6 [8.83 to 25.47] | 0.7 [0.00 to 5.06] | 0.5 [0.00 to 4.76] | 0.0 [0.0 to 3.69]

15. Secondary Outcome: Median Calculated Annualized Bleeding Rate for Treated Target Joint Bleeds
Description: as for outcome 14
Time Frame: From Baseline to at least 24 weeks
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Median (Inter-Quartile Range); unit: Treated target joint bleeds per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 14 | 29 | 27 | 15
Treated target joint bleeds per year | 6.5 [0.00 to 19.68] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 1.13] | 0.0 [0.00 to 0.00]

16. Secondary Outcome: Intra-Participant Comparison of the Calculated Annualized Bleeding Rate for Treated Bleeds With Emicizumab Prophylaxis On-Study Versus With Previous Episodic Therapy Pre-Study
Description: This is an intra-participant comparison of the annualized bleeding rate (ABR) for treated bleeds pre-study versus on-study in the non-interventional study (NIS) population previously treated with episodic therapy in NIS BH29768. The number of treated bleeds over the efficacy period is presented here as a calculated ABR that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated bleed was defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: Efficacy periods: At least 24 weeks prior to study entry (mean [min-max] for A+B NIS-Previous Episodic Therapy: 183 [169-221] days); and From Baseline to at least 24 weeks on study (mean [min-max] for A+B NIS-Emicizumab: 363 [324-422] days)
Population: A total of 4 participants, pooled from Arm A and Arm B (2 per Arm), who participated in the NIS BH29768 before entering this study were included for this intraparticipant analysis.
Measure: Mean (Full Range); unit: Treated bleeds per year
Groups:
- A+B NIS: Previous Episodic Therapy Pre-Study: Only participants with hemophilia A (with or without FVIII inhibitors), pooled from Arm A and Arm B, who previously participated in the NIS BH29768 are included here for analysis. This previous episodic therapy analysis group includes historical bleed data during participation in NIS BH29768 prior to enrollment in this study from 2 patients enrolled in Arm A who had FVIII inhibitors and had received episodic therapy with bypassing agents and 2 patients enrolled in Arm B who did not have FVIII inhibitors and had received episodic therapy with FVIII.
- A+B NIS: Emicizumab Prophylaxis On-Study: Only participants with hemophilia A (with or without FVIII inhibitors), pooled from Arm A and Arm B, who previously participated in the NIS BH29768 are included here for analysis. On this study, the participants received prophylactic emicizumab at a dose of 3 mg/kg via SC injection QW for the first 4 weeks, followed by either 1.5 mg/kg (in Arm A) or 6 mg/kg (in Arm B) via SC injection Q4W for at least 24 weeks. After 24 weeks of treatment, participants were allowed to continue receiving emicizumab until marketing authorization, as part of this study or a separate extension study, as long as they derived clinical benefit. Participants continued to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
Arm/Group | A+B NIS: Previous Episodic Therapy Pre-Study | A+B NIS: Emicizumab Prophylaxis On-Study
Number analyzed (Participants) | 4 | 4
Treated bleeds per year | 13.02 [4.96 to 21.61] | 0.24 [0.00 to 0.97]

17. Secondary Outcome: Intra-Participant Comparison of the Calculated Annualized Bleeding Rate for All Bleeds With Emicizumab Prophylaxis On-Study Versus With Previous Episodic Therapy Pre-Study
Description: This is an intra-participant comparison of the annualized bleeding rate (ABR) for all bleeds pre-study versus on-study in the non-interventional study (NIS) population previously treated with episodic therapy in NIS BH29768. The ABR was calculated for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. All bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. "All bleeds" comprises both treated and non-treated bleeds, and the 72-hour rule was implemented separately for each type. For treated bleeds, the 72-hour rule meant that two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. For non-treated bleeds, the 72-hour rule was calculated as a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Full Range); unit: All bleeds per year
Arm/Group | A+B NIS: Previous Episodic Therapy Pre-Study | A+B NIS: Emicizumab Prophylaxis On-Study
Number analyzed (Participants) | 4 | 4
All bleeds per year | 39.67 [15.13 to 92.55] | 2.04 [1.10 to 3.38]

18. Secondary Outcome: Arms A, B, and C: Adjusted Mean Hemophilia A Quality of Life (Haem-A-QoL) Questionnaire Physical Health Domain Score at Week 25 in Participants ≥18 Years of Age
Description: The Haem-A-QoL questionnaire has been developed and used in hemophilia A participants, assessing very specific aspects of dealing with hemophilia. The questionnaire consists of items pertaining to 10 domains: physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feeling, relationships, treatment, view of yourself, and outlook for the future. The total score for each domain ranges from 0 to 100 with lower scores reflective of better quality of life. Physical Health domain score is reported (range 0 to 100, with lower scores reflective of better physical health). The means were derived via an analysis of covariance (ANCOVA) model and have been adjusted for the following co-variates: baseline score, treatment group, and treatment by baseline interaction term.
Time Frame: Baseline and Week 25
Population: Adult participants randomized to Arms A, B, and C. The number analyzed represents participants who provided responses at Baseline and Week 25.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W
Number analyzed (Participants) | 8 | 25 | 21
score on a scale | 42.53 (14.00) | 27.85 (19.82) | 24.20 (16.09)
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW; Test type: Superiority; p = 0.0515, ANCOVA — Type I error controlled; Means were adjusted for baseline score, treatment group, and treatment by baseline interaction term; Difference in Adjusted Means = 14.68, 95% CI 2-sided [-0.10 to 29.46] — The difference in adjusted means was calculated as Arm C minus Arm A
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W; Test type: Superiority; p = 0.0204, ANCOVA — Type I error controlled; Means were adjusted for baseline score, treatment group, and treatment by baseline interaction term; Difference in Adjusted Means = 18.33, 95% CI 2-sided [2.97 to 33.68] — The difference in adjusted means was calculated as Arm C minus Arm B

19. Secondary Outcome: Arms A, B, and C: Change From Baseline to Week 25 in Haem-A-QoL Questionnaire Physical Health Domain Score for Participants ≥18 Years of Age
Description: The Haem-A-QoL questionnaire has been developed and used in hemophilia A participants, assessing very specific aspects of dealing with hemophilia. The questionnaire consists of items pertaining to 10 domains: physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feeling, relationships, treatment, view of yourself, and outlook for the future. The total score for each domain ranges from 0 to 100 with lower scores reflective of better quality of life. Physical Health domain score is reported (range 0 to 100, with lower scores reflective of better physical health).
Time Frame: Baseline and Week 25
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W
Number analyzed (Participants) | 8 | 25 | 21
score on a scale
  Absolute Value at Baseline (BL) | 51.25 (23.41) | 50.60 (20.38) | 42.14 (14.10)
  Change from BL to Week 25 | -5.63 (14.00) | -20.20 (19.82) | -22.14 (16.09)

20. Secondary Outcome: Arms A, B, and C: Adjusted Mean Haem-A-QoL Questionnaire Total Score at Week 25 in Participants ≥18 Years of Age
Description: The Haem-A-QoL questionnaire has been developed and used in hemophilia A participants, assessing very specific aspects of dealing with hemophilia. The questionnaire consists of items pertaining to 10 domains: physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feeling, relationships, treatment, view of yourself, and outlook for the future. The total score for each domain ranges from 0 to 100 with lower scores reflective of better quality of life. Haem-A-QoL Total Score is the average of all domain scores and it ranges from 0 to 100, with lower scores reflective of better quality of life. The means were derived via an analysis of covariance (ANCOVA) model and have been adjusted for the following co-variates: baseline score, treatment group, and treatment by baseline interaction term.
Time Frame: Baseline and Week 25
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W
Number analyzed (Participants) | 8 | 25 | 21
score on a scale | 43.32 (7.47) | 37.26 (16.17) | 29.30 (14.60)
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW; Test type: Superiority; p = 0.3281, ANCOVA — Not controlled for Type I error; Means were adjusted for baseline score, treatment group, and treatment by baseline interaction term; Difference in Adjusted Means = 6.06, 95% CI 2-sided [-6.27 to 18.40] — The difference in adjusted means was calculated as Arm C minus Arm A
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W; Test type: Superiority; p = 0.0297, ANCOVA — Not controlled for Type I error; Means were adjusted for baseline score, treatment group, and treatment by baseline interaction term; Difference in Adjusted Means = 14.01, 95% CI 2-sided [1.44 to 26.59] — The difference in adjusted means was calculated as Arm C minus Arm B

21. Secondary Outcome: Arms A, B, and C: Change From Baseline to Week 25 in Haem-A-QoL Questionnaire Total Score for Participants ≥18 Years of Age
Description: The Haem-A-QoL questionnaire has been developed and used in hemophilia A participants, assessing very specific aspects of dealing with hemophilia. The questionnaire consists of items pertaining to 10 domains: physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feeling, relationships, treatment, view of yourself, and outlook for the future. The total score for each domain ranges from 0 to 100 with lower scores reflective of better quality of life. Haem-A-QoL Total Score is the average of all domain scores and it ranges from 0 to 100, with lower scores reflective of better quality of life.
Time Frame: Baseline and Week 25
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W
Number analyzed (Participants) | 8 | 25 | 21
score on a scale
  Value at Baseline (BL) | 42.05 (17.89) | 49.15 (16.04) | 46.59 (12.58)
  Change from BL to Week 25 | -2.50 (7.47) | -10.14 (16.17) | -17.61 (14.60)

22. Secondary Outcome: Arms A, B, and C: Hemophilia-Specific Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Total Score at Baseline and Week 25 in Participants 12 to 17 Years of Age
Description: The Haemo-QoL-SF contains 35 items covering nine dimensions considered relevant for the adolescent's (aged 12-17 years) health-related quality of life (HRQoL). Items are rated with five respective response options: never, seldom, sometimes, often, and always. The score ranges from 0 to 100, and a higher score is indicative of poorer HRQoL. According to the pre-specified statistical analysis plan, no statistical analyses were performed on the protocol-defined endpoints for the Haemo-QoL-SF due to the small number of adolescents randomized to Arms A, B and C.
Time Frame: Baseline and Week 25
Population: Only adolescents (aged 12-17 years) randomized to Arms A, B, and C were included in this analysis. The number analyzed represents participants who provided responses at Baseline and Week 25.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W
Number analyzed (Participants) | 2 | 3 | 5
score on a scale
  Value at Baseline (BL) | 44.7 [35.0 to 54.3] | 44.5 [35.7 to 58.6] | 35.7 [20.0 to 50.7]
  Value at Week 25 | 21.5 [13.6 to 29.3] | 32.9 [27.9 to 39.3] | 27.6 [10.0 to 40.0]

23. Secondary Outcome: Arms A, B, and C: Adjusted Mean European Quality of Life 5-Dimensions-5 Levels Questionnaire (EQ-5D-5L) Questionnaire Visual Analog Scale (VAS) Score at Week 25
Description: EQ-5D-5L is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L VAS. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. The means were derived via an analysis of covariance (ANCOVA) model and have been adjusted for the following co-variates: baseline score, treatment group, and treatment by baseline interaction term.
Time Frame: Baseline and Week 25
Population: Participants randomized to Arms A, B, and C. The number analyzed represents participants who provided responses at Baseline and Week 25.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W
Number analyzed (Participants) | 9 | 28 | 25
score on a scale | 78.36 (20.68) | 81.82 (23.19) | 85.94 (15.20)
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW; Test type: Superiority; p = 0.6165, ANCOVA — Not controlled for Type I error; Means were adjusted for baseline score, treatment group, and treatment by baseline interaction term; Difference in Adjusted Means = -3.46, 95% CI 2-sided [-17.23 to 10.31] — The difference in adjusted means was calculated as Arm C minus Arm A
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W; Test type: Superiority; p = 0.2797, ANCOVA — Not controlled for Type I error; Means were adjusted for baseline score, treatment group, and treatment by baseline interaction term; Difference in Adjusted Means = -7.58, 95% CI 2-sided [-21.48 to 6.33] — The difference in adjusted means was calculated as Arm C minus Arm B

24. Secondary Outcome: Arms A, B, and C: Change From Baseline in EQ-5D-5L Questionnaire VAS Score at Week 25
Description: The European Quality of Life 5-Dimensions-5 Levels Questionnaire (EQ-5D-5L) is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L VAS. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Baseline and Week 25
Population: The number analyzed indicates the number of participants who responded to the questionnaire scale at a given timepoint. For the change from baseline analysis, only participants who responded at both Baseline and Week 25 were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W
Number analyzed (Participants) | 10 | 29 | 25
score on a scale
  Value at Baseline (BL) | 84.50 (15.07) | 74.59 (16.91) | 78.96 (12.91)
  Change from BL to Week 25: number analyzed (Participants) | 9 | 28 | 25
  Change from BL to Week 25 | -2.00 (13.27) | 4.82 (19.13) | 7.40 (16.67)

25. Secondary Outcome: Arms A, B, and C: Adjusted Mean EQ-5D-5L Index Utility Score at Week 25
Description: The European Quality of Life 5-Dimensions-5 Levels Questionnaire (EQ-5D-5L) is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L VAS. The EQ-5D-5L health state profile is designed to record the participant's current health state in 5 domains: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression. Responses from the five domains are used to calculate a single index utility score on a scale of 0 to 1, with higher scores reflective of better quality of life. The means were derived via an analysis of covariance (ANCOVA) model and have been adjusted for the following co-variates: baseline score, treatment group, and treatment by baseline interaction term.
Time Frame: Baseline and Week 25
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W
Number analyzed (Participants) | 9 | 28 | 25
score on a scale | 0.74 (0.35) | 0.79 (0.27) | 0.82 (0.17)
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW; Test type: Superiority; p = 0.4890, ANCOVA — Not controlled for Type I error; Means were adjusted for baseline score, treatment group, and treatment by baseline interaction term; Difference in Adjusted Means = -0.05, 95% CI 2-sided [-0.18 to 0.09] — The difference in adjusted means was calculated as Arm C minus Arm A
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W; Test type: Superiority; p = 0.2454, ANCOVA — Not controlled for Type I error; Means were adjusted for baseline score, treatment group, and treatment by baseline interaction term; Difference in Adjusted Means = -0.08, 95% CI 2-sided [-0.22 to 0.06] — The difference in adjusted means was calculated as Arm C minus Arm B

26. Secondary Outcome: Arms A, B, and C: Change From Baseline in EQ-5D-5L Index Utility Score at Week 25
Description: The European Quality of Life 5-Dimensions-5 Levels Questionnaire (EQ-5D-5L) is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L VAS. The EQ-5D-5L health state profile is designed to record the participant's current health state in 5 domains: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression. Responses from the five domains are used to calculate a single index utility score on a scale of 0 to 1, with higher scores reflective of better quality of life.
Time Frame: Baseline and Week 25
Population: Participants randomized to Arms A, B, and C. The number analyzed indicates the number of participants who responded to the questionnaire scale at a given timepoint. For the change from baseline analysis, only participants who responded at both Baseline and Week 25 were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W
Number analyzed (Participants) | 10 | 29 | 25
score on a scale
  Value at Baseline (BL) | 0.76 (0.27) | 0.68 (0.27) | 0.75 (0.20)
  Change from BL to Week 25: number analyzed (Participants) | 9 | 28 | 25
  Change from BL to Week 25 | 0.02 (0.09) | 0.08 (0.22) | 0.08 (0.21)

27. Secondary Outcome: Arm D: Change From Baseline in Haemo-QoL-SF Questionnaire Physical Health and Total Scores at Week 25 in Participants 8 to 12 Years of Age
Description: The Hemophilia-Specific Quality of Life Short Form (Haemo-QoL-SF) questionnaire contains 35 items covering nine dimensions considered relevant for the children's health-related quality of life (HRQoL). Items are rated with five respective response options: never, seldom, sometimes, often, and always. The scores range from 0 to 100, and higher scores are indicative of poorer HRQoL.
Time Frame: Baseline and Week 25
Population: This outcome measure was only applicable for participants enrolled in Arm D. The number analyzed for each visit represents the number of participants who responded to the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
Number analyzed (Participants) | 6
score on a scale
  Physical Health Score: Baseline (BL) - Value at Visit | 67.71 (30.98)
  Physical Health Score: Change from BL at Week 25: number analyzed (Participants) | 5
  Physical Health Score: Change from BL at Week 25 | -53.75 (37.66)
  Total Score: Baseline (BL) Value at Visit | 54.40 (19.68)
  Total Score: Change from BL at Week 25: number analyzed (Participants) | 5
  Total Score: Change from BL at Week 25 | -23.86 (17.84)

28. Secondary Outcome: Arm D: Change From Baseline in the Caregiver-Reported Adapted Health-Related Quality of Life for Hemophilia Patients With Inhibitors (Adapted Inhib-QoL) Including Aspects of Caregiver Burden Questionnaire Score Over Time
Description: Proxy assessment of HRQoL and aspects of caregiver burden for all children, regardless of age, were collected using the Adapted Inhib-QoL with Aspects of Caregiver Burden questionnaire. The questionnaire comprises two parts. The first part asks the caregiver for his/her opinion on the child's HRQoL (proxy HRQoL). The second part asks the caregiver to rate how the child's situation is for them (i.e., the impact of the child's disease and treatment on the caregiver). Items are rated with 5 respective response options: never, seldom, sometimes, often, and all the time. Scores range from 0 to 100, with lower scores reflective of better HRQoL. A total score is calculated as the sum of all of the items in the scale.
Time Frame: Baseline (Week 1) and Weeks 17, 29, 37, and 49, every 12 weeks during extension phase, and study completion (up to 48 months)
Reporting Status: Not Posted, anticipated posting 2026-05

29. Secondary Outcome: Number of Participants With Adverse Events by Severity, According to the World Health Organization (WHO) Toxicity Grading Scale
Time Frame: From Baseline until end of study (up to 85 months)
Reporting Status: Not Posted

30. Secondary Outcome: Number of Participants With Adverse Events Leading to Study Drug Discontinuation
Time Frame: From Baseline until end of study (up to 85 months)
Reporting Status: Not Posted

31. Secondary Outcome: Number of Participants With Thromboembolic Events by Severity, According to the WHO Toxicity Grading Scale
Time Frame: From Baseline until end of study (up to 85 months)
Reporting Status: Not Posted

32. Secondary Outcome: Number of Participants With Thrombotic Microangiopathy by Severity, According to the WHO Toxicity Grading Scale
Time Frame: From Baseline until end of study (up to 85 months)
Reporting Status: Not Posted

33. Secondary Outcome: Number of Participants With Injection-Site Reactions by Severity, According to the WHO Toxicity Grading Scale
Time Frame: From Baseline until end of study (up to 85 months)
Reporting Status: Not Posted

34. Secondary Outcome: Number of Participants With Severe Hypersensitivity, Anaphylaxis, or Anaphylactoid Reactions
Time Frame: From Baseline until end of study (up to 85 months)
Reporting Status: Not Posted

35. Secondary Outcome: Number of Participants With Serum Chemistry Laboratory Abnormalities by Highest WHO Grade Post-Baseline, According to the WHO Toxicity Grading Scale
Time Frame: From Baseline until end of study (up to 85 months)
Reporting Status: Not Posted

36. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities by Highest WHO Grade Post-Baseline, According to the WHO Toxicity Grading Scale
Time Frame: From Baseline until end of study (up to 85 months)
Reporting Status: Not Posted

37. Secondary Outcome: Change From Baseline in Body Temperature Over Time
Time Frame: Baseline, Weeks 5, 25, 49, and at study completion (up to 85 months)
Reporting Status: Not Posted

38. Secondary Outcome: Change From Baseline in Pulse Rate Over Time
Time Frame: Baseline, Weeks 5, 25, 49, and at study completion (up to 85 months)
Reporting Status: Not Posted

39. Secondary Outcome: Change From Baseline in Respiratory Rate Over Time
Time Frame: Baseline, Weeks 5, 25, 49, and at study completion (up to 85 months)
Reporting Status: Not Posted

40. Secondary Outcome: Change From Baseline in Systolic Blood Pressure Over Time
Time Frame: Baseline, Weeks 5, 25, 49, and at study completion (up to 85 months)
Reporting Status: Not Posted

41. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure Over Time
Time Frame: Baseline, Weeks 5, 25, 49, and at study completion (up to 85 months)
Reporting Status: Not Posted

42. Secondary Outcome: Number of Participants With Anti-Emicizumab Antibodies
Time Frame: QW: Pre-dose at Weeks 1, 5, 9, 13, 17, 21, 25, 33, 41, 49, and every 12 weeks thereafter until study completion; Q4W: Pre-dose at Weeks 1, 5, 9, 13, 17, 21, 25, and every 12 weeks thereafter until study completion (up to 85 months)
Reporting Status: Not Posted

43. Secondary Outcome: Plasma Trough Concentration (Ctrough) of Emicizumab
Time Frame: QW: Predose at Weeks 1, 2, 3, 4, 5, 7, 9, 13, 17, 21, 25, 33, 41, 49, and every 12 weeks thereafter to study completion; Q4W: Predose at Weeks 1, 2, 3, 4, 5, 7, 9, 13, 17, 21, 25, and every 12 weeks thereafter to study completion (up to 85 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the date of randomization or enrollment until the clinical cutoff date (Arms A to C: Emicizumab, up to 223 weeks; Arm D: up to 67 weeks; Arm C [Control] No Prophylaxis: up to 28 weeks)
Description: The study is ongoing and adverse event data are still being collected. These results will be updated within 1 year of the final data collection date (i.e., the last patient's last visit).
Groups:
- Arm C (Emi): 6 mg/kg Emicizumab Prophylaxis Q4W: After 24 weeks on no prophylaxis, participants were given the opportunity to switch to receive emicizumab prophylaxis at 3 mg/kg QW via SC injection for 4 weeks, followed by 6 mg/kg Q4W until marketing authorization as part of this study or a separate extension study, as long as they derive clinical benefit. Participants continued to receive standard-of-care treatments on an episodic basis for the treatment of breakthrough bleeds during the study.
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W | Arm C (Emi): 6 mg/kg Emicizumab Prophylaxis Q4W | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/29 | 0/27 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 8/29 | 4/27 | 2/14 | 0/15
Other Adverse Events (participants affected / at risk) | 2/14 | 27/29 | 24/27 | 11/14 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C (Control): No Prophylaxis (N=14) | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW (N=29) | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W (N=27) | Arm C (Emi): 6 mg/kg Emicizumab Prophylaxis Q4W (N=14) | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW (N=15)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C (Control): No Prophylaxis (N=14) | Arm A: 1.5 mg/kg Emicizumab Prophylaxis QW (N=29) | Arm B: 6 mg/kg Emicizumab Prophylaxis Q4W (N=27) | Arm C (Emi): 6 mg/kg Emicizumab Prophylaxis Q4W (N=14) | Arm D: 1.5 mg/kg Emicizumab Prophylaxis QW (N=15)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 11 (17) | 10 (22) | 8 (16) | 6 (21)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (5) | 3 (3) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (7) | 6 (10) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5) | 5 (10) | 3 (7) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (8)
Blood glucose increased (Investigations) | 0 (0) | 3 (7) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood ketone body increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Differential white blood cell count abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (6) | 2 (2) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 4 (7) | 5 (29) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (7) | 1 (1) | 0 (0) | 3 (4)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (8) | 4 (4) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (3) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 5 (5) | 2 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (3)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palipitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-04-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03315455/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03315455/SAP_001.pdf